CLINICAL TRIAL: NCT04872504
Title: Performance of the Hypotension Prediction Index With Invasive Arterial Pressure Waveform in Liver Transplantation
Brief Title: Hypotension Prediction Index in Patients Undergoing Liver Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Hypotension prediction index
Record Dates: First submitted 2021-04-26; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Intraoperative Hypotension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Acumen HPI-enabled EV1000 screen (Experimental): Acumen HPI-enabled EV1000 screen
  Interventions: Device: Acumen HPI-enabled EV1000 screen

INTERVENTIONS:
Device: Acumen HPI-enabled EV1000 screen — Acumen HPI-enabled EV1000 screen record the incidence of intraoperative hypotension

SUMMARY:
A prospective, open-label and single-center study to determine whether the use of Acumen Hypotension Prediction Index software predicts the occurrence of hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥ 20 years;
* Scheduled liver transplantation
* Planned pressure monitoring with an arterial line;
* General anesthesia

Exclusion Criteria:

* Contraindication for invasive blood pressure monitoring
* End-staged renal disease
* pre-operative MAP <65 mmHg
* Severe heart failure
* Severe cardiac shunt
* Severe aortic stenosis
* Severe atrial fibrillation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Accurate hypotension prediction of EV1000 system | MAP measurements of each case were recorded every 20 s by the EV1000 system from induction to the end of surgery, assessed up to 1 day.
  Analyze the actual incidence of hypotension after HPI alarm more than 85 within 15 min
Incidence of intraoperative hypotension | MAP measurements of each case were recorded every 20 s by the EV1000 system from induction to the end of surgery, assessed up to 1 day
  Frequency, duration of intraoperative hypotension, which defined as MAP < 65 mmHg at least 1 min
Severity of intraoperative hypotension | MAP measurements of each case were recorded every 20 s by the EV1000 system from induction to the end of surgery, assessed up to 1 day
  MAP measurements were recorded every 20 s by the EV1000 system from induction to Time-weighted average mean arterial pressure (TWA-MAP) < 65 mmHg

SECONDARY OUTCOMES:
Hospital stay and ICU stay | Days from admission to discharge, assessed up to 1 month
  The incidence and severity of intraoperative hypotension correlate with patient's hospital stay and ICU stay
Mortality after surgery | Days from admission to discharge, assessed up to 1 month
  The incidence and severity of intraoperative hypotension correlate with patient's mortality
Adverse effects | Days from admission to discharge, assessed up to 1 month
  The incidence and severity of hypotension correlate with the adverse effects like acute liver failure, acute kidney injury and acute myocardial injury

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No